CLINICAL TRIAL: NCT01702532
Title: A Study to Evaluate Relief of Provoked Acute Craving by Nicotine Mouth Film and Nicotine Lozenge
Brief Title: Nicotine Mouth Film for Craving Relief.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RH01589
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Smoking Cessation
Keywords: provoked craving
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Mouth Film (Experimental): mint nicotine mouth film, buccal administration
  Interventions: Drug: Nicotine
- Nicotine Lozenge (Active Comparator): nicotine lozenge, buccal administration
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Comparison of different dosage forms of nicotine

SUMMARY:
Nicotine mouth film is a new dosage form of nicotine replacement therapy. The purpose of this study is to investigate the craving relief efficacy of nicotine mouth film by comparing mint nicotine mouth film to nicotine lozenge in light smokers using the provoked craving model. The cues used to provoke a craving episode will be the sight and smell of a lit cigarette and the manipulations required to light a cigarette. The smokers will be denied access to cigarettes for 4 hours prior to the provoked craving session in order to precipitate nicotine withdrawal and an increase level of cigarette craving.

ELIGIBILITY:
Inclusion Criteria:

* BMI within the range of 19-35 kg/m2;
* Current cigarette smokers who have smoked regularly daily for at least a year,
* Participants who smoke their first cigarette more than 30 minutes after waking up

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity to nicotine (or closely related compounds) or any of the stated ingredients in formulation.
* Any participant whose CO level rises during the sequestration period (i.e., the subject's two expired CO assessments immediately prior to the provoked craving paradigm are higher than the mean baseline CO assessment) and, in the opinion of the investigator, may have smoked during that time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Los Angeles Clinical Trials, Burbank, California
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: A total of 386 participants were screened of which 322 subjects were randomized into the study. Sixty subjects were screen failures, Two subjects withdrew consent and an additional 2 subjects were not randomized due to other reasons.
Groups:
- Nicotine Mouth Film 2.5 mg: Participants received a single dose of 2.5 mg nicotine mouth film placed on the top of tongue and pressed to the roof of mouth until film dissolved (approximately 2 to 3 minutes).
- Nicotine Lozenge 2 mg: Participants received a single dose of 2 mg nicotine lozenge to be placed into the mouth and periodically moved from one side of mouth to other, without swallowing until lozenge dissolved (approximately 20 to 30 minutes).
Period: Overall Study
Arm/Group | Nicotine Mouth Film 2.5 mg | Nicotine Lozenge 2 mg
Started | 161 | 161
Safety Population | 161 | 160 (One subject randomized but did not receive the study treatment.)
Completed | 161 | 160
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Lozenge 2 mg: Participants received a single dose of 2 mg nicotine lozenge to be placed into the mouth and periodically moved from one side of mouth to other, without swallowing until lozenge dissolved (approximately 20 - 30 minutes).
- Total: Total of all reporting groups
Arm/Group | Nicotine Mouth Film 2.5 mg | Nicotine Lozenge 2 mg | Total
Number analyzed (Participants) | 161 | 160 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (12.91) | 39.8 (12.64) | 39.4 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 73 | 162
  Male | 72 | 87 | 159

OUTCOME MEASURES:

1. Primary Outcome: The Change From Pre-dose Post-provocation in Craving Score at 50 Seconds
Description: Participants completed a cigarette craving assessment consisting of the following five items: "I have a desire for a cigarette right now; If it were possible I would smoke right now; All I want right now is a cigarette; I have an urge for a cigarette; I crave a cigarette right now. All participants indicated craving intensity on a pre-drawn 100 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 (disagree) to 100 (agree). The average of the scores over the five items was defined as craving score for each time point.
Time Frame: Pre-dosing post-provocation to 50 seconds
Population: All randomized participants who took at least one dose of medication and provided at least one valid craving assessment measurement on-treatment. Any participant with a missing response to any of the five craving assessment items was considered as a missing value and was imputed.
Measure: Least Squares Mean (Inter-Quartile Range); unit: mm
Arm/Group | Nicotine Mouth Film 2.5 mg | Nicotine Lozenge 2 mg
Number analyzed (Participants) | 161 | 160
mm | -14.15 [-16.90 to -11.41] | -9.26 [-12.01 to -6.50]
Statistical Analysis 1: Comparison: Nicotine Mouth Film 2.5 mg vs Nicotine Lozenge 2 mg; Null hypotheses considered change in craving score means from pre-dose post-provocation at 50 seconds to be equal for the two treatment groups; Test type: Superiority or Other; p = 0.0141, ANCOVA — The comparison between treatments was conducted in a hierarchical order; consequently no adjustment of the significance level (5%) for multiplicity was needed; ANCOVA model contains pre-provocation baseline, pre-dosing post-provocation craving score, and the terms treatment groups and center as fixed; LS Means Difference = -4.90, 95% CI 2-sided [-8.80 to -0.99] — Comment: The confidence interval is for the difference between treatments groups

2. Secondary Outcome: The Change From Pre-dose Post-provocation in Craving Score at 3, 5, 7, 10, 15, 20, 25, and 30 Minutes
Description: Participants completed a cigarette craving assessment consisting of the following five items: "I have a desire for a cigarette right now; If it were possible I would smoke right now; All I want right now is a cigarette; I have an urge for a cigarette; I crave a cigarette right now. All participants indicated craving intensity on a pre-drawn 100 mm VAS ranging from 0 (disagree) to 100 (agree). The average of the scores over the five items was defined as the craving score for each time .
Time Frame: Pre-dosing post-provocation to 3, 5, 7, 10, 15, 20, 25, and 30 minutes
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Nicotine Mouth Film 2.5 mg | Nicotine Lozenge 2 mg
Number analyzed (Participants) | 161 | 160
mm
  Difference in VAS Score at 3 Minutes | -27.02 [-30.64 to -23.39] | -20.30 [-23.93 to -16.67]
  Difference in VAS Score at 5 Minutes | -33.95 [-37.88 to -30.02] | -28.33 [-32.27 to -24.38]
  Difference in VAS Score at 7 Minutes | -39.13 [-43.20 to -35.05] | -34.14 [-38.23 to -30.05]
  Difference in VAS Score at 10 Minutes | -40.94 [-45.08 to -36.80] | -39.16 [-43.31 to -35.01]
  Difference in VAS Score at 15 Minutes | -42.19 [-46.42 to -37.97] | -42.30 [-46.53 to -38.06]
  Difference in VAS Score at 20 Minutes | -42.43 [-46.77 to -38.09] | -45.23 [-49.58 to -40.87]
  Difference in VAS Score at 25 Minutes | -43.16 [-47.55 to -38.78] | -46.27 [-50.67 to -41.88]
  Difference in VAS Score at 30 Minutes | -43.54 [-48.11 to -38.97] | -47.48 [-52.06 to -42.89]

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of the sequestration period upto 5 days after the last treament
Arm/Group | Nicotine Mouth Film 2.5 mg | Nicotine Lozenge 2 mg
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/160
Other Adverse Events (participants affected / at risk) | 6/161 | 29/160
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Mouth Film 2.5 mg (N=161) | Nicotine Lozenge 2 mg (N=160)
Nausea (Gastrointestinal disorders) | 1 (1) | 14 (14)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.